CLINICAL TRIAL: NCT04482530
Title: Food Matrices Based on Fruit Pastes as Vectors of Carbohydrates for the Prevention and Management of Protein-energy Undernutrition in the Elderly: Proof of Clinical Concept
Brief Title: Food Matrices Based on Fruit Pastes as Vectors of Carbohydrates for the Prevention and Management of Protein-energy Undernutrition in the Elderly (Fruisenior)
Acronym: Fruisenior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unité de Nutrition Humaine, INRAE, Centre Auvergne-Rhône Alpes (Unknown); Unité de recherche CSGA, INRAE Dijon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: RBHP 2019 PICKERING; 2019-A00995-52 (Other: ANSM)
Record Dates: First submitted 2020-06-16; First posted 2020-07-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Fruit pastes matrices; Elderly healthy volunteer; Dietary intake

STUDY DESIGN:
Who Masked: Participant
Masking Description: Same flavor will be used for all matrices. The different matrices will be offered to volunteers in in individual packaged portions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Original recipe (Experimental): Normal fruit paste
  Interventions: Other: fruit paste matrice
- maltodextrin recipe (Experimental): fruit pastes in which some of the simple sugars in the recipe will be replaced by maltodextrin with a low glycemic index (DE12).
  Interventions: Other: fruit paste matrice
- fructose recipe (Experimental): fruit pastes in which some of the simple sugars in the recipe (25% min) will be replaced by fructose
  Interventions: Other: fruit paste matrice
- isomaltulose recipe (Experimental): fruit pastes with some of the sugars will be replaced (25% min) by isomaltulose
  Interventions: Other: fruit paste matrice
- mixed recipe (Experimental): fruit pastes with some of the sugars will be replaced (25% min) by fructose / isomaltulose
  Interventions: Other: fruit paste matrice

INTERVENTIONS:
Other: fruit paste matrice — Evaluation of the kinetics of the appearance of nutrients and the metabolic response induced by the consumption of fruit pastes (5 different matrices will be tested: 1 Original recipe, 1 maltodextrine recipe, 1 fructose recipe, 1 isomaltulose recipe and 1 mixed recipe comprising fructose and isomaltulose) in elderly healthy volunteers.

SUMMARY:
To develop more natural fruit pastes matrices that can effectively act as carbohydrate vectors in the elderly population and that are part of a normal diet while maintaining the pleasure of eating.

DETAILED DESCRIPTION:
This is an interventional randomized, single blinded, cross over and controlled study.

The main objective is the study of the kinetic modification of blood glucose with the "fruit" matrices enriched in maltodextrins, fructose and isomaltulose compared to the original recipe consisting only of simple sugars.

The secondary objective is:

-the assessment of the acceptability of all the fruit pastes tested (organoleptic, satiety and gastrointestinal comfort aspects).The study is composed of 7 visits Visit 1 - Selection Visit (Day -7)

* Informed consent form
* Clinical examination
* Medical history
* Anthropometric characteristics
* Blood biochemical and hematological assessment
* Compliance test with the original matrix will be carried out

Visit 2 (D0) / Visit 3 (D7) / Visit 4 (D14) / Visit 5 (D21) / Visit 6 (D28): study period If all the biological criteria are respected, the subjects will have to come back to the clinical center for each of the 5 study periods.

Volunteers will arrive fasted, without smoking in the morning. A catheter will be placed for blood sampling. After a first blood sampling for basal values, volunteers will ingest the equivalent of two bars of fruit pastes (about 80g in 10 minutes maximum) and blood will be withdrawn 15, 30, 45, 60, 90, 120 and 180 minutes after ingestion. The different matrices (5 in total) will be tested on the same volunteer. Plasma samples will be used to determine plasma glucose and fructose concentrations (aliquots stored in center for later assays) to evaluate the postprandial profiles of these two nutrients. At the end of the kinetic, the volunteers will be offered a complete meal. A satiety questionnaire will be performed before then 60 and 180 min after the ingestion of each fruit matrix. A questionnaire of satisfaction and acceptability will also be realized during the consumption of the matrix.

After the 5 fruit matrix will be tested, the subject will be invited to participate in an individual interview of about 30-45min with a member of the project team. The purpose of this interview will be a qualitative approach to search for a food development that can could improve the sensory quality of the fruit pastes tested and intended for the elderly (see below).

Visit 7 (D35 to D40): Participation in a discussion group (about 2 hours). During the participation in this group all 10 participants will be invited to taste the 5 products (original recipe, maltodextrin recipe, fructose recipe, isomaltulose recipe and mixed recipe comprising fructose and isomaltulose). Participants will be asked to indicate for each product their degree of appreciation for these products, their possible defects and qualities and to suggest ideas for improving their taste / texture / appearance. These interviews will alternate individual reflection phases and discussion phases according to the focus group method.

Visit 7 will be the last visit of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male subject
* Subject over 65 years (included)
* Subject over 61 kg (included)
* Able to consume the 80g of fruit pastes in 10 minutes
* Subject with a dentition consistent with the fruit paste consumption in 10 minutes
* Subject with a Body Mass Index (BMI) between 21 and 30 kg/m2
* Subject agreeing to provide written consent

Exclusion Criteria:

* Subject with acute pathology (unstable or terminal pathology, severe dementia)
* Subject with renal failure (clearance < 60 ml/min)
* Subject with metabolic syndrome (3 of the following 5 criteria: waist greater than 94 cm, blood triglyceride greater than 1.7 mmol/l, blood pressure greater than or equal to 130 mm Hg/85 mm Hg, cholesterol (HDL) less than 1.0 mmol/l in men, blood glucose greater than or equal to 5.6 mmol/l)
* Person with diabetes
* Subject on food restriction
* Subject undergoing chemotherapy
* Subject with gastrointestinal pathology
* Subject in a diet incompatible with the nutritional protocol (gluten, lactose or milk intolerance, vegan)

Min Age: 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-31 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve (AUC) of glycemia | Day 0
  Area Under the Curve (AUC) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glycemia | Day 0
  Maximum Plasma Concentration (Cmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glycemia | Day 0
  Time of Maximum Plasma Concentration (Tmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glycemia | Day 7
  Area Under the Curve (AUC) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glycemia | Day 7
  Maximum Plasma Concentration (Cmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glycemia | day 7
  Time of Maximum Plasma Concentration (Tmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glycemia | day 14
  Area Under the Curve (AUC) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glycemia | day 14
  Maximum Plasma Concentration (Cmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glycemia | day 14
  Time of Maximum Plasma Concentration (Tmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glycemia | day 21
  Area Under the Curve (AUC) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glycemia | day 21
  Maximum Plasma Concentration (Cmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glycemia | day 21
  Time of Maximum Plasma Concentration (Tmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glycemia | day 28
  Area Under the Curve (AUC) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glycemia | day 28
  Maximum Plasma Concentration (Cmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of glycemia | day 28
  Time of Maximum Plasma Concentration (Tmax) of glycemia (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) of fructose | Day 0
  Area Under the Curve (AUC) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of fructose | Day 0
  Maximum Plasma Concentration (Cmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of fructose | Day 0
  Time of Maximum Plasma Concentration (Tmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of fructose | Day 7
  Area Under the Curve (AUC) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of fructose | Day 7
  Maximum Plasma Concentration (Cmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of fructose | Day 7
  Time of Maximum Plasma Concentration (Tmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of fructose | Day 14
  Area Under the Curve (AUC) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of fructose | Day 14
  Maximum Plasma Concentration (Cmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of fructose | Day 14
  Time of Maximum Plasma Concentration (Tmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of fructose | Day 21
  Area Under the Curve (AUC) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of fructose | Day 21
  Maximum Plasma Concentration (Cmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of fructose | Day 21
  Time of Maximum Plasma Concentration (Tmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of fructose | Day 28
  Area Under the Curve (AUC) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of fructose | Day 28
  Maximum Plasma Concentration (Cmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of fructose | Day 28
  Time of Maximum Plasma Concentration (Tmax) of fructose (defined in g/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glucagon | day 0
  Area Under the Curve (AUC) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glucagon | day 0
  : Maximum Plasma Concentration (Cmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glucagon | day 0
  Time of Maximum Plasma Concentration (Tmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glucagon | day 7
  Area Under the Curve (AUC) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of glucagon | day 7
  Maximum Plasma Concentration (Cmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of glucagon | Day 7
  Time of Maximum Plasma Concentration (Tmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of glucagon | Day 14
  Area Under the Curve (AUC) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of glucagon | Day 14
  Maximum Plasma Concentration (Cmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glucagon | Day 14
  Time of Maximum Plasma Concentration (Tmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of glucagon | Day 21
  Area Under the Curve (AUC) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of glucagon | Day 21
  Maximum Plasma Concentration (Cmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glucagon | Day 21
  Time of Maximum Plasma Concentration (Tmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of glucagon | Day 28
  Area Under the Curve (AUC) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of glucagon | Day 28
  Maximum Plasma Concentration (Cmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of glucagon | Day 28
  Time of Maximum Plasma Concentration (Tmax) of glucagon (defined in np/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of CCK | Day 0
  Area Under the Curve (AUC) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of CCK | Day 0
  Maximum Plasma Concentration (Cmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of CCK | Day 0
  Time of Maximum Plasma Concentration (Tmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of CCK | Day 7
  Area Under the Curve (AUC) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of CCK | Day 7
  Maximum Plasma Concentration (Cmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of CCK | Day 7
  Time of Maximum Plasma Concentration (Tmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of CCK | Day 14
  Area Under the Curve (AUC) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of CCK | Day 14
  Maximum Plasma Concentration (Cmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of CCK | Day 14
  Time of Maximum Plasma Concentration (Tmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of CCK | Day 21
  Area Under the Curve (AUC) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of CCK | Day 21
  Maximum Plasma Concentration (Cmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of CCK | Day 21
  Time of Maximum Plasma Concentration (Tmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of CCK | Day 28
  Area Under the Curve (AUC) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of CCK | Day 28
  Maximum Plasma Concentration (Cmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of CCK | Day 28
  Time of Maximum Plasma Concentration (Tmax) of CCK (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of Grehlin | Day 0
  Area Under the Curve (AUC) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of Grehlin | Day 0
  Maximum Plasma Concentration (Cmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of Grehlin | day 0
  Time of Maximum Plasma Concentration (Tmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of Grehlin | day 7
  Area Under the Curve (AUC) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of Grehlin | day 7
  Maximum Plasma Concentration (Cmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of Grehlin | day 7
  Time of Maximum Plasma Concentration (Tmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of Grehlin | day 14
  Area Under the Curve (AUC) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of Grehlin | day 14
  Maximum Plasma Concentration (Cmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of Grehlin | day 14
  Time of Maximum Plasma Concentration (Tmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of Grehlin | day 21
  Area Under the Curve (AUC) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of Grehlin | day 21
  Maximum Plasma Concentration (Cmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of Grehlin | day 21
  Time of Maximum Plasma Concentration (Tmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of Grehlin | day 28
  Area Under the Curve (AUC) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of Grehlin | day 28
  Maximum Plasma Concentration (Cmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of Grehlin | day 28
  Time of Maximum Plasma Concentration (Tmax) of Grehlin (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of leptin | day 0
  Area Under the Curve (AUC) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of leptin | day 0
  Maximum Plasma Concentration (Cmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of leptin | day 0
  Time of Maximum Plasma Concentration (Tmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of leptin | day 7
  Area Under the Curve (AUC) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of leptin | day 7
  Maximum Plasma Concentration (Cmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of leptin | day 7
  Time of Maximum Plasma Concentration (Tmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of leptin | day 14
  Area Under the Curve (AUC) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of leptin | day 14
  Maximum Plasma Concentration (Cmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of leptin | day 14
  Time of Maximum Plasma Concentration (Tmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of leptin | day 21
  Area Under the Curve (AUC) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of leptin | day 21
  Maximum Plasma Concentration (Cmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of leptin | day 21
  Time of Maximum Plasma Concentration (Tmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of leptin | day 28
  Area Under the Curve (AUC) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of leptin | day 28
  Maximum Plasma Concentration (Cmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of leptin | day 28
  Time of Maximum Plasma Concentration (Tmax) of leptin (defined in ng/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of GLP1 | day 0
  Area Under the Curve (AUC) of GLP1 (defined in pmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of GLP1 | day 0
  Maximum Plasma Concentration (Cmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of GLP1 | day 0
  Time of Maximum Plasma Concentration (Tmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of GLP1 | day 7
  Area Under the Curve (AUC) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of GLP1 | day 7
  Maximum Plasma Concentration (Cmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of GLP1 | day 7
  Time of Maximum Plasma Concentration (Tmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of GLP1 | day 14
  Area Under the Curve (AUC) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of GLP1 | day 14
  Maximum Plasma Concentration (Cmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of GLP1 | day 14
  Time of Maximum Plasma Concentration (Tmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of GLP1 | day 21
  Area Under the Curve (AUC) of GLP1 (defined in pmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of GLP1 | day 21
  Maximum Plasma Concentration (Cmax) of GLP1 (defined in pmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of GLP1 | day 21
  Time of Maximum Plasma Concentration (Tmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of GLP1 | day 28
  Area Under the Curve (AUC) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of GLP1 | day 28
  Maximum Plasma Concentration (Cmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of GLP1 | day 28
  Time of Maximum Plasma Concentration (Tmax) of GLP1 (defined in pmol /L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of incretines | day 0
  Area Under the Curve (AUC) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of incretines | day 0
  Maximum Plasma Concentration (Cmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of incretines | day 0
  Time of Maximum Plasma Concentration (Tmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of incretines | day 7
  Area Under the Curve (AUC) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of incretines | day 7
  Maximum Plasma Concentration (Cmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of incretines | day 7
  Time of Maximum Plasma Concentration (Tmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of incretines | day 14
  Area Under the Curve (AUC) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of incretines | day 14
  Maximum Plasma Concentration (Cmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of incretines | day 14
  Time of Maximum Plasma Concentration (Tmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of incretines | day 21
  Area Under the Curve (AUC) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of incretines | day 21
  Maximum Plasma Concentration (Cmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of incretines | day 21
  Time of Maximum Plasma Concentration (Tmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of incretines | day 28
  Area Under the Curve (AUC) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of incretines | day 28
  Maximum Plasma Concentration (Cmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of incretines | day 28
  Time of Maximum Plasma Concentration (Tmax) of incretines (defined in pg/mL) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of insulin | day 0
  Area Under the Curve (AUC) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of insulin | day 0
  Maximum Plasma Concentration (Cmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of insulin | day 0
  Time of Maximum Plasma Concentration (Tmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of insulin | day 7
  Area Under the Curve (AUC) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of insulin | day 7
  Maximum Plasma Concentration (Cmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of insulin | day 7
  Time of Maximum Plasma Concentration (Tmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of insulin | day 14
  Area Under the Curve (AUC) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of insulin | day 14
  Maximum Plasma Concentration (Cmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of insulin | day 14
  Time of Maximum Plasma Concentration (Tmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Area Under the Curve (AUC) of insulin | day 21
  Area Under the Curve (AUC) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of insulin | day 21
  Maximum Plasma Concentration (Cmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of insulin | day 21
  Time of Maximum Plasma Concentration (Tmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of insulin | day 28
  Area Under the Curve (AUC) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of urea | day 28
  Maximum Plasma Concentration (Cmax) of urea (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of insulin | day 28
  Time of Maximum Plasma Concentration (Tmax) of insulin (defined in µg/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of urea | day 0
  Area Under the Curve (AUC) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of urea | day 0
  Maximum Plasma Concentration (Cmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of urea | day 0
  Time of Maximum Plasma Concentration (Tmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of urea | day 7
  Area Under the Curve (AUC) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of urea | day 7
  Maximum Plasma Concentration (Cmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of urea | day 7
  Time of Maximum Plasma Concentration (Tmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of urea | day 14
  Area Under the Curve (AUC) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Maximum Plasma Concentration (Cmax) of urea | day 14
  Maximum Plasma Concentration (Cmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of urea | day 14
  Time of Maximum Plasma Concentration (Tmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of urea | day 21
  Area Under the Curve (AUC) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of urea | day 21
  Maximum Plasma Concentration (Cmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Time of Maximum Plasma Concentration (Tmax) of urea | day 21
  Time of Maximum Plasma Concentration (Tmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Area Under the Curve (AUC) of urea | day 28
  Area Under the Curve (AUC) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Maximum Plasma Concentration (Cmax) of urea | day 28
  Maximum Plasma Concentration (Cmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste.
Time of Maximum Plasma Concentration (Tmax) of urea | day 28
  Time of Maximum Plasma Concentration (Tmax) of urea (defined in mmol/L) between T0 and T120 minutes following ingestion of fruit paste
Questionnaire of satiety | at time 0 after ingestion in Day 0
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 60 after ingestion in Day 0
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry
Questionnaire of satiety | at time 180 after ingestion in Day 0
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 0 after ingestion in Day 7
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry
Questionnaire of satiety | at time 60 after ingestion in Day 7
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry
Questionnaire of satiety | at time 180 after ingestion in Day 7
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 0 after ingestion in Day 14
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 60 after ingestion in Day 14
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry
Questionnaire of satiety | at time 180 after ingestion in Day 14
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry
Questionnaire of satiety | at time 0 after ingestion in Day 21
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 60 after ingestion in Day 21
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 180 after ingestion in Day 21
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 0 after ingestion in Day 28
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 60 after ingestion in Day 28
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of satiety | at time 180 after ingestion in Day 28
  Questionnaire was composed of 4 questions where satiety was assessed by a 0-10 Numerical Satiety Rating Scale where "0" means to be free from hunger and "10" to be very hungry.
Questionnaire of acceptability | day 0
  Acceptability was assessed by a 7-point time scale where "1" means a very poor acceptability and "7" means a very good acceptability
Questionnaire of acceptability | day 7
  Acceptability was assessed by a 7-point time scale where "1" means a very poor acceptability and "7" means a very good acceptability
Questionnaire of acceptability | day 14
  Acceptability was assessed by a 7-point time scale where "1" means a very poor acceptability and "7" means a very good acceptability
Questionnaire of acceptability | day 21
  Acceptability was assessed by a 7-point time scale where "1" means a very poor acceptability and "7" means a very good acceptability
Questionnaire of acceptability | day 28
  Acceptability was assessed by a 7-point time scale where "1" means a very poor acceptability and "7" means a very good acceptability
Facilited individual interview | day 40
  Facilitated interview to assess organoleptic, satiety and gastrointestinal comfort
Focus group | day 40
  Focus group interview to assess organoleptic, satiety and gastrointestinal comfort

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle Pickering, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France